CLINICAL TRIAL: NCT04995471
Title: Comparing the Effectiveness of Telerehabilitation vs. in Presence Rehabilitation of Reading Disorders, Using a Rhythm-based Intervention for Reading (Rhythmic Reading Training, RRT)
Brief Title: Telerehabilitation vs. in Presence Rehabilitation of Reading Disorders Using the Rhythmic Reading Training (RRT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Alice Cancer, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRT vs. RRTT
Record Dates: First submitted 2021-07-16; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Developmental Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- In presence RRT - prototype software (Experimental): 10 biweekly in presence sessions of 45 minutes supervised by a trainer
  Interventions: Behavioral: In presence RRT - prototype software
- In presence RRT - online platform (Experimental): 10 biweekly in presence sessions of 45 minutes supervised by a trainer
  Interventions: Behavioral: In presence RRT - online platform
- Tele-RRT - prototype software (Experimental): 10 biweekly telerehabilitation sessions of 45 minutes supervised by a trainer
  Interventions: Behavioral: Tele-RRT - prototype software
- Tele-RRT - online platform (Experimental): 10 biweekly telerehabilitation sessions of 45 minutes supervised by a trainer
  Interventions: Behavioral: Tele-RRT - online platform
- No intervention (No Intervention): 5 weeks no intervention period

INTERVENTIONS:
Behavioral: In presence RRT - prototype software — Rhythmic Reading Training (RRT) is a prototype software which includes reading exercises presented simultaneously with a rhythmic stimulation with gradually increasing speed.
  Arms: In presence RRT - prototype software
Behavioral: In presence RRT - online platform — RRT is a web application with a client-server structure developed in javascript/php language using open-source support libraries. The server-side system uses a LAMP stack (Linux, Apache, Mysql, Php) on Server Cloud. The application can also be activated as a desktop application through "portable web server" installation systems, available for linux, windows and OS operating systems. In this form, the application can also be used in contexts without an Internet connection. The system is also accessible from tablets. RRT consists of a module of progressive reading exercises. The exercises are organized according to different types (syllables, words, non-words, short texts) and accompanied by a rhythmic-melodic stimulation, which is coordinated with a visual cue. Both remote (Rhythmic Reading Tele-Training, RRTT) and in presence administration (RRT) are available.
  Arms: In presence RRT - online platform
Behavioral: Tele-RRT - prototype software — Rhythmic Reading Training (RRT) is a prototype software which includes reading exercises presented simultaneously with a rhythmic stimulation with gradually increasing speed.
  Arms: Tele-RRT - prototype software
Behavioral: Tele-RRT - online platform — RRT is a web application with a client-server structure developed in javascript/php language using open-source support libraries. The server-side system uses a LAMP stack (Linux, Apache, Mysql, Php) on Server Cloud. The application can also be activated as a desktop application through "portable web server" installation systems, available for linux, windows and OS operating systems. In this form, the application can also be used in contexts without an Internet connection. The system is also accessible from tablets. RRT consists of a module of progressive reading exercises. The exercises are organized according to different types (syllables, words, non-words, short texts) and accompanied by a rhythmic-melodic stimulation, which is coordinated with a visual cue. Both remote (Rhythmic Reading Tele-Training, RRTT) and in presence administration (RRT) are available.
  Arms: Tele-RRT - online platform

SUMMARY:
The aim of the study is to compare the effectiveness of telerehabilitation vs. in presence rehabilitation of reading disorders, using a rhythm-based intervention for reading (i.e., Rhythmic Reading Training)

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with DD (ICD-10 code: F81.0) on the basis of standard inclusion and exclusion criteria (ICD-10: World Health Organization, 1992) and of the diagnosis procedure followed in the Italian practice

Exclusion Criteria:

* presence of comorbidity with other neuropsychiatric or psychopathological conditions
* having been involved in previous reading intervention programs in the previous 3 months

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Word reading - DDE-2 | 5 weeks
  Word reading speed in syllable / seconds
Word reading - DDE-2 | 5 weeks
  Word reading accuracy in n. of errors
Word reading - DDE-2 | 3 months
  Word reading speed in syllable / seconds
Word reading - DDE-2 | 3 months
  Word reading accuracy in n. of errors
Pseudo-word reading - DDE-2 | 5 weeks
  Pseudo-word reading speed in syllable / seconds
Pseudo-word reading - DDE-2 | 5 weeks
  Pseudo-word reading accuracy in n. of errors
Pseudo-word reading - DDE-2 | 3 months
  Pseudo-word reading speed in syllable / seconds
Pseudo-word reading - DDE-2 | 3 months
  Pseudo-word reading accuracy in n. of errors
Text reading - MT-3-Clinica Battery | 5 weeks
  Text reading speed in syllable / seconds
Text reading - MT-3-Clinica Battery | 5 weeks
  Text reading accuracy in n. of errors
Text reading - MT-3-Clinica Battery | 3 months
  Text reading speed in syllable / seconds
Text reading - MT-3-Clinica Battery | 3 months
  Text reading accuracy in n. of errors

SECONDARY OUTCOMES:
Phonemic awareness task (Judica et al., in press) | 5 weeks
  N. of errors in phonemic blending + N. of errors phonemic elision
Phonemic awareness task (Judica et al., in press) | 3 months
  N. of errors in phonemic blending + N. of errors phonemic elision
Digit span (Wechsler Intelligence Scale for Children-IV, WISC-IV) | 5 weeks
  Forward and backward digit span
Digit span (Wechsler Intelligence Scale for Children-IV, WISC-IV) | 3 months
  Forward and backward digit span
Rapid Automatized naming task - RAN (De Luca et al., 2005) | 5 weeks
  RAN Speed in seconds
Rapid Automatized naming task - RAN (De Luca et al., 2005) | 3 months
  RAN Speed in seconds
Rhythm reproduction task | 5 weeks
  N. of correctly reproduced rhythmic patterns
Rhythm reproduction task | 3 months
  N. of correctly reproduced rhythmic patterns

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cancer A, Sarti D, De Salvatore M, Granocchio E, Chieffo DPR, Antonietti A. Dyslexia Telerehabilitation during the COVID-19 Pandemic: Results of a Rhythm-Based Intervention for Reading. Children (Basel). 2021 Nov 5;8(11):1011. doi: 10.3390/children8111011. PMID 34828724